CLINICAL TRIAL: NCT06132815
Title: The Efficacy of Different Gingival Displacement Methods Before Definitive Digital Impression: A Randomized Controlled Clinical Trial
Brief Title: The Efficacy of Different Gingival Displacement Methods Before Definitive Digital Impression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Elashry, Assistant Lecturer of Fixed Prosthodontics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: #2/2022
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Gingival Displacement
MeSH Terms: interventions — Astringents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Laser troughing (Experimental)
  Interventions: Device: Laser troughing
- Retraction cord and astringent (Experimental)
  Interventions: Other: Retraction cord and astringent
- Cordless retraction paste with astringent (Experimental)
  Interventions: Other: Cordless retraction paste with astringent
- Cordless retraction paste without astringent (Active Comparator)
  Interventions: Other: Cordless retraction paste without astringent

INTERVENTIONS:
Device: Laser troughing — Laser troughing will be carried out by passing laser optic fiber in contact mode along the gingival sulcus. Laser energy will be delivered with a wavelength of 980nm and power of 0.8W, in continuous mode. Laser tip will be inserted 1mm into the gingival sulcus, to facilitate an accurate recording of finish line
  Arms: Laser troughing
Other: Retraction cord and astringent — Partial isolation of the tooth with cotton rolls and saliva ejector will be performed. Appropriate size of retraction cord will be soaked in astringent for 5 mins. Then packing of the cord will be started from the mesial interproximal area by gently packing into the sulcus with the gingival cord packer instrument using the single cord technique. Retraction cord will be kept in place for 5 minutes. Cord will be removed immediately before the start of the intraoral scan
  Arms: Retraction cord and astringent
Other: Cordless retraction paste with astringent — The cordless paste with astringent will be injected gently into the sulcus, leaning on the tooth at the point of the cervical limit and not on the gingiva, the cannula will remain parallel to the axis of the tooth to exert optimal pressure. Then it will removed after 5 mins with copiously irrigated water until no traces of the materials left.
  Arms: Cordless retraction paste with astringent
Other: Cordless retraction paste without astringent — The cordless paste without astringent 10 will be injected into the sulcus of the gingiva. The suitable size of Comprecap will be held on the abutment to push the material deep into the sulcus of the gingiva, and the participants will be informed to bite over it for a period of 3 to 5 minutes. After 5 minutes, the comprecap with the set retraction material attached to it, will be removed from the patient mouth.
  Arms: Cordless retraction paste without astringent

SUMMARY:
This study aims to evaluate and compare the efficacy of four methods in achieving vertical and horizontal gingival tissue displacement to be captured by optical digital impression. Moreover, the effect of the gingival displacement methods on the periodontal tissues around the final restoration will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients having normal occlusion.
* Good oral hygiene with no signs of periapical pathology or periodontal disease (plaque index score ≤10).
* Clinically and radiographically healthy gingiva and periodontium around the abutments with no evidence of attachment loss.
* Thick gingival biotype (determination using color coded probe).
* Patient having natural teeth as opposing dentition.
* Gingival sulcus of the abutment teeth (≤ 3mm).
* Adequate abutment tooth length for retention without deep subgingival extension (not more than 0.5mm)

Exclusion Criteria:

* Pregnancy, which prevents the use of diagnostic x-rays.
* Parafunctional habits.
* Mobility of abutment teeth.
* Gingival Recession
* Patient presenting allergy to materials being used.
* Smoking.
* Medical history that could affect their periodontal condition.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Horizontal displacement measurement | up to one month
  All measurements were obtained from the definitive digital impression by using dental intraoral scanner software. Horizontal displacement was measured as the distance from the most prominent point of the crest of the marginal gingiva to the finish line in the same crowns section (in the same plane).
Vertical Displacement measurement | up to one month
  All measurements were obtained from the definitive digital impression by using dental intraoral scanner software. Vertical displacement will be measured as the distance from the most prominent point of the finish line to the deepest point of gingival sulcus.

SECONDARY OUTCOMES:
Dental plaque measurement | up to one month
  Using the plaque index of Silness and Loe. Each tooth will be scored from 0-3 according to the amount of plaque accumulation.
  0: No plaque in the gingival area.
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
Gingival inflammation measurement | up to one month
  Using the gingival index of Silness and Loe. Each tooth will be scored from 0-3 according to the degree of gingival inflammation.
  0: Normal gingiva
  1. Mild inflammation - slight change in color, slight oedema. No bleeding on probing
  2. Moderate inflammation-redness, oedema and glazing. Bleeding on probing
  3. Severe inflammation - marked redness and oedema. Ulceration. Tendency to spontaneous bleeding
Gingival Height loss measurement | up to one month
  Complete arch maxillary digital impressions (postoperative scans) will be made for each patient by using intraoral scanner after cementation of the crowns. The postoperative scans will be superimposed by the pre-operative scan. A cross sectional line will be drawn in the middle of the superimposed scans and the measurements will be done at 2 points (midbuccal and midlingual). The distance from the gingival margin of the preoperative scan to that of one postoperative scan will be considered gingival height loss at the scan's timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Elashry, MSc, Principal Investigator — Alexandria University; Sanaa Hussein, PhD, Study Chair — Alexandria University; Ihab Hammad, PhD, Study Chair — Alexandria University; Rania Fahmy, PhD, Study Chair — Alexandria University; Islam M Abdel Raheem, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt